CLINICAL TRIAL: NCT02834104
Title: Validation of Fibrosis Quantification Using T1 Mapping Against Histology as Reference and Comparison With Fibrosis Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-30; 2011-A01395-36 (Other: ansm)
Record Dates: First submitted 2016-07-05; First posted 2016-07-15 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Fibrosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myocardial fibrosis (Experimental)
  Interventions: Device: RMI; Other: myocardial biopsy; Biological: blood sample

INTERVENTIONS:
Device: RMI
Other: myocardial biopsy
Biological: blood sample

SUMMARY:
Myocardial fibrosis is recognized as the pathologic entity of extracellular matrix remodeling. Diffuse, reactive fibrosis is increasingly recognized in a variety of conditions despite the absence of ischemia. Regardless of the etiology, fibrosis leads to increased myocardial stiffness thereby promoting cardiac dysfunction. This dysfunction may present clinically with symptoms of cardiac failure although this is often a subclinical disease. Various imaging modalities and collagen biomarkers have been used as surrogate markers to assess the presence, extent, and turnover of myocardial fibrosis. Techniques using echocardiography, cardiac magnetic resonance, and nuclear imaging have been developed to detect early features of systolic and diastolic left ventricular dysfunction and impaired contractile reserve. Further identification of diffuse reactive fibrosis may be possible with evolving cardiac magnetic resonance and molecular techniques. The goal of this protocol is to validate cardiac magnetic resonance imaging as a new tool for fibrosis quantification against histology as standard of reference.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require surgical aortic valve replacement , which will benefit from an MRI to measure fibrosis in the months preceding the surgery.
* Patient submitted to the social security scheme
* Patient agreeing to participate in the study and who signed the informed consent.

Exclusion Criteria:

* A history of myocardial
* Unstable Patients requiring treatment with catecholamines.
* hepatocellular insufficiency of alcoholic origin
* Severe renal impairment
* Appearance before examining coronary syndrome at high risk, defined according to international recommendations.
* History of known allergy to gadolinium at diagnosis
* Pregnant or lactating
* Patient < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11-18 (Actual); Primary Completion 2015-12-19 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
quantification of myocardial fibrosis by RMI | 5years

SECONDARY OUTCOMES:
measuring biomarkers of fibrosis | 5 years
  BLOOD SAMPLE

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided